CLINICAL TRIAL: NCT04895306
Title: Exploring the Role of Testosterone as a Novel Anti-Nociceptive Agent in Women With Chronic Pain and Opioid Use
Brief Title: Testosterone Replacement to Alleviate Pain in Postmenopausal Women (TRAPP Trial)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Shehzad Basaria, M.D., Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021P001447
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Pain; Opioid Use; Androgen Deficiency; Back Pain
Keywords: Opioid Use; Pain; Women; Testosterone; Back Pain
MeSH Terms: conditions — Pain; Back Pain | interventions — testosterone 17 beta-cypionate; Testosterone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Testosterone (Experimental): Weekly intramuscular administration at a dose of 3 mg
  Interventions: Drug: Testosterone Cypionate
- Placebo (Placebo Comparator): Weekly intramuscular administration of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Testosterone Cypionate — Weekly intramuscular administration of testosterone at a dose of 3 mg
  Other Names: testosterone
  Arms: Testosterone
Drug: Placebo — Weekly intramuscular administration of Placebo
  Arms: Placebo

SUMMARY:
The aim of this trial is to evaluate whether testosterone replacement results in greater improvement in pain perception, pain tolerance, sexual function, physical function and quality of life when compared with placebo in women with chronic back pain treated with opioids who have low testosterone.

DETAILED DESCRIPTION:
This single-center, randomized, double-blind, placebo-controlled, parallel-group trial will evaluate pain and quality of life outcomes associated with 3 months of treatment with testosterone or placebo in women aged 60 years or older with chronic non-cancer back pain who are taking opioid analgesics for at least 6 months and have low testosterone.

ELIGIBILITY:
Inclusion Criteria:

* Women, age 60 years and older.
* Chronic non-cancer back pain.
* Use of opioid analgesics for at least 6 months.
* Serum total testosterone <8.7 ng/dL and/or free testosterone <0.47 pg/mL.
* Normal mammogram within the last 12 months
* Endometrial thickness of <4 mm in women with an intact uterus assessed by endometrial ultrasound.
* Ability and willingness to provide informed consent.

Exclusion Criteria:

* History of breast or endometrial cancer
* Estrogen therapy in the past 3 months
* Baseline hematocrit >48%.
* Serum creatinine >2.5 mg/dL.
* HbA1c >9.0%. Subjects on insulin therapy will be excluded.
* BMI >40 kg/m2.
* Uncontrolled congestive heart failure.
* Myocardial infarction, acute coronary syndrome, revascularization surgery or stroke within the past 3 months.
* History of genetic thromboembolic disorder.
* Diagnosis of bipolar disorder or schizophrenia.
* Use of testosterone, spironolactone, finasteride or systemic ketoconazole in the past 3 months.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain Interference Subscale score of the Brief Pain Inventory (BPI) questionnaire | 3 months
  The Pain Interference Subscale of the BPI is specifically relevant to patients with chronic back pain who are using opioids and correlates strongly with the patient's quality of life.

SECONDARY OUTCOMES:
Algometer-induced Pressure Pain | 3 months
  A digital pressure algometer at the trapezius muscle and the metacarpophalangeal joint of the thumb was used to measure pressure pain thresholds. Higher values represent a better tolerance of pressure pain.
Weighted Pinprick Stimulator-induced Mechanical Pain | 3 months
  Weighted pinprick stimulators are used to assess mechanical pain. Lower values represent better tolerance of pain
Ice Water-induced Cold Pain and Its After-sensation | 3 months
  Cold-pressor tests measure cold-induced pain and its sensation. Time was measured when a participant reached pain tolerance in cold water and after sensation. Higher values of time in Cold pain tolerance and lower values of time in Cold pain after-sensation (30 seconds) represent better tolerance of pain.
Health Quality of Life (QoL) as Assessed by Short Form 36 (SF-36) | 3 months
  The SF-36 measures 8 domains of the QoL: physical function, bodily pain, vitality, role limitations due to physical problems, general health perceptions, emotional well-being, social function, and role limitations due to emotional problems. Each domain is scored separately from 0 to 100 with higher scores representing better health-related QoL.
Mood and well-being, assessed using the by Positive and Negative Affect Scale (PANAS) affectivity balance scale | 3 months
  The PANAS affectivity balance scale includes 10 questions evaluating positive and negative affect.
Physical function, assessed using the 6-minute walk test (6-MWT) | 3 months
  Subjects will be asked to walk for 6 minutes at a comfortable pace on a premeasured flat surface; gait speed will be calculated by the distance walked (m) in 6 minutes. The 6-minute walk test (6-MWT) is an objective test of physical function validated in older adults and in women with chronic low back pain.
Sexual Function assessed by the Female Sexual Distress Scale (FSDS) | 3 months
  For this 13-item questionnaire, women rate each item in terms of frequency from 0 (never) to 4 (always). Items are summed to create a total score ranging from 0 to 52, with higher scores indicating more sexually related distress

CONTACTS AND LOCATIONS:
Overall Officials: Shehzad Basaria, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States